CLINICAL TRIAL: NCT01859910
Title: Compression of the Lid Margin Increase Microbial Contamination Risk of Patients Undergoing Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orbis (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Tiantian Ye, Zhongshan Ophthalmic Center, Orbis
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: Lid margin VS Cataract Surgery
Record Dates: First submitted 2013-05-20; First posted 2013-05-22 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- compression (Experimental): compression and scrub of lid margin for 5 circles before cataract surgery
  Interventions: Procedure: compression and scrub of lid margin; Procedure: routine preparation for cataract
- control (Active Comparator): no compression or scrub of lid margin
  Interventions: Procedure: routine preparation for cataract

INTERVENTIONS:
Procedure: compression and scrub of lid margin — compression and scrub of lid margin for 5 circles before cataract surgery
  Arms: compression
Procedure: routine preparation for cataract

SUMMARY:
To investigate whether compression of the lid margin increase microbial contamination risk of patients undergoing cataract surgery

ELIGIBILITY:
Inclusion Criteria:

* (1) Age > 60 years; (2) clinical diagnosis of age related cataract, without previous recent ocular surgery; (3) undergoing phacoemulsification with implantation of intraocular lens ; (4) able to give informed consent.

Exclusion Criteria:

* (1) any inflammation of the eye or other parts of the body within the previous 3 months; (2) chronic use of any types ophthalmic medication; (3) contact lens wear; (4) ocular surgery within the past 3 months; (5) use of systemic antibiotics within 30 days; (6) use of eyedrops in either eye within 3 days of enrollment; (7) need for concurrent glaucoma, cornea or other surgery.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2011-10; Primary Completion 2012-04 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
positive rate of culture | 5months

SECONDARY OUTCOMES:
bacteria distribution of the culture | 5months

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China